CLINICAL TRIAL: NCT05151913
Title: Exploratory, Prospective, Non-therapeutic, Paired- Matched Controlled Two-arm Study to Investigate the Microbiome Composition in Women With Recurring Intrahepatic Cholestasis of Pregnancy (ICP)
Brief Title: The Microbiome Composition in Women With Recurring Intrahepatic Cholestasis of Pregnancy (ICP)
Status: Completed | Type: Observational
Sponsor: MetaboGen AB (Industry)
Collaborators: Skane University Hospital (Other); Stockholm South General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: META001
Record Dates: First submitted 2021-10-25; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Intrahepatic Cholestasis of Pregnancy
Keywords: Pregnancy; Microbiome
MeSH Terms: conditions — Intrahepatic Cholestasis of Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal samples are collected for analyzing the gut microbiome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Previous ICP, recurrence: Pregnant women with at least one previously completed parturition with ICP and ICP during the present study
  Interventions: Other: Exploratory
- Previous ICP, non-recurrence: Pregnant women with at least one previously completed parturition with ICP and no ICP during the present study
  Interventions: Other: Exploratory
- No previous ICP: Pregnant women with at least one previously completed parturition with no previous ICP and no ICP during the present study
  Interventions: Other: Exploratory

INTERVENTIONS:
Other: Exploratory — Fecal microbiome

SUMMARY:
This is an exploratory non-therapeutic study to study the microbiome patterns during pregnancy in women with ICP in order to identify specific bacterial strains for further product development.

DETAILED DESCRIPTION:
Intrahepatic Cholestasis in Pregnancy (ICP) is a disease that appears in the later stage of pregnancy with itching (pruritus) and increased risk of fetal complications. It is the most prevalent pregnancy-specific liver disease, affecting between 1 and 20 % of all pregnant women, depending on ethnicity and geographic location.

The condition is associated with an increased risk of adverse fetal outcomes, including preterm labour and intrauterine death. Further, ICP is associated with an increased risk for pre-eclampsia, thyroid disease, diabetes and cancer. ICP is typically present during the third trimester, when the serum concentrations of progesterone and estrogens reach their peak, and also, the time when the gut barrier has an increased permeability. In ICP subjects, both altered progesterone and bile acid metabolism is observed.

The underlying etiology for ICP is unknown, but there are indications that the gut microbiota may be involved. It has become increasingly clear that the gut microbiota is associated with metabolic diseases and has an important function in metabolizing endogenous and dietary metabolites. Bile acids are metabolized by the gut microbiota by deconjugation and production of secondary metabolites, ursodeoxycholic acid (UDCA) being one example of a secondary bile acid produced by the microbiota. Bile acids are produced from cholesterol by a series of hepatic enzymes generating cholic acid (CA) and chenodeoxycholic acid (CDCA) in humans that are conjugated to predominantly glycine. These primary bile acids are stored in the gall bladder from where they are released upon a meal. The majority of conjugated bile acids are reabsorbed from the ileum, but through the action of microbial bile salt hydrolase (BSH), the bile acids escape reabsorption and enter the colon where they can be further metabolized. Accordingly, bile acid deconjugation reduces enterohepatic recirculation of bile acids and thereby reduces the total bile acid pool. Reduction of bile acid levels are crucial to reduce pruritus and reduce fetal complication risks in ICP.

The aim is to identify biomarkers in the microbiota associated with ICP and the onset of this disease, or state of the disease, during pregnancy. Bacterial species that have a capability for UDCA production and correlate with sulphated progesterone metabolites are of specific interest. Furthermore, bacteria with sulphating and desulphating capabilities are also of interest.

ELIGIBILITY:
Inclusion Criteria:

Arm 1

* Pregnant woman > 18 years
* Signed informed consent for participation
* At least one previously completed parturition with ICP
* Willingness and ability to comply with the study procedures, visit schedules and other instructions regarding the study

Arm 2

* Pregnant woman ≥ 18 years (±5 calendar years from the matched subject in arm 1)
* Signed informed consent for participation
* At least one previously completed parturition
* No previous ICP
* Willingness and ability to comply with the study procedures, visit schedules and other instructions regarding the study

Exclusion Criteria:

* Multifetal pregnancy (twins, triplets etc.)
* Latin American ethnicity
* Use of any systemic antibiotics within 3 months prior to enrollment
* Medical history of liver disease (other than previous ICP for subjects in arm 1)
* Medically significant gastrointestinal disorder which, in the opinion of the investigator, may affect the results or the subject ́s ability to comply with the study
* History or concurrent status of any clinically significant disease or disorder which, in the opinion of the investigator, may influence the results or the subject ́s ability to participate in the study
* Participation in any other clinical study that included drug treatment within 3 months prior to enrollment
* Serious bacterial or chronic viral infection such as human immunodeficiency virus (HIV) or hepatitis virus at enrollment visit
* Any other condition which, in the Investigator ́s opinion, makes the subject unsuitable for study participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women with previous ICP and matched controls
Study Population: Pregnant women with previously completed parturition with intrahepatic cholestasis of pregnancy and matched controls
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2019-10-14 (Actual)

PRIMARY OUTCOMES:
Gut microbiome composition | Pregnancy week 9+0 - 19+6 until 6 weeks post-partum (+ 2 weeks)
  Change in gut microbiome composition

SECONDARY OUTCOMES:
Bile acids levels | Pregnancy week 9+0 - 19+6 until 6 weeks post-partum (+ 2 weeks)
  Change in total and individual bile acids
Liver function test AST | Pregnancy week 9+0 - 19+6 until 6 weeks post-partum (+ 2 weeks)
  Change in AST
Liver function test ALT | Pregnancy week 9+0 - 19+6 until 6 weeks post-partum (+ 2 weeks)
  Change in ALT
Liver function test GGT | Pregnancy week 9+0 - 19+6 until 6 weeks post-partum (+ 2 weeks)
  Change in GGT
Liver function test bilirubin | Pregnancy week 9+0 - 19+6 until 6 weeks post-partum (+ 2 weeks)
  Change in bilirubin

CONTACTS AND LOCATIONS:
Overall Officials: Helena Strevens, MD, PhD, Principal Investigator — Skane University Hospital, Sweden
Locations (2):
- Sweden (2):
  - Skane University Hospotal, Lund
  - Stockholm South General Hospital, Stockholm